CLINICAL TRIAL: NCT05710900
Title: DECIDE: DiEt ChoIce to Promote Type 2 Diabetes REmission Supported by Community Pharmacists and Registered Dietitians
Brief Title: DiEt ChoIce to Promote Type 2 Diabetes REmission
Acronym: DECIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H22-03055
Record Dates: First submitted 2023-01-16; First posted 2023-02-02 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: low-carbohydrate diets; low-calorie diets; type 2 diabetes remission
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Pilot implementation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-calorie diet group (Experimental): A low-calorie diet involving will involve a commercial weight loss program (pre-packaged foods from Ideal Protein, select lean protein sources, non-starchy vegetables) and be led by the pharmacist and registered dietitian (RD) involving in-person and virtual appointments.
  Interventions: Other: Dietary intervention
- Low-carbohydrate diet group (Experimental): The low-carbohydrate diet will involve an individualized whole-food diet (30-130 grams carbohydrate per day) led through virtual visits with a registered dietitian.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Each dietary remission strategy involves three phases focused on weight loss and medication deprescribing (Phase 1: Weeks 0-12), transition to an individualized sustainable dietary pattern (Phase 2: Weeks 13-20), and weight loss/remission maintenance (Phase 3: Weeks 21-52).

SUMMARY:
Type 2 diabetes is typically viewed as a chronic, progressive, and lifelong condition. Patients and their healthcare providers "manage" type 2 diabetes through lifestyle modifications and various types of medications designed to lower blood sugar.

Exciting new research indicates that "remission" of type 2 diabetes - defined as returning blood sugar into the normal range without having to use medications - through therapeutic nutrition may be possible for many people living with the condition.

We will examine the preference, adherence and clinical results of a low-calorie diet or low-carbohydrate diet in type 2 diabetes remission rates.

DETAILED DESCRIPTION:
Each dietary remission strategy involves three phases focused on weight loss and medication deprescribing (Phase 1: Weeks 0-12), transition to an individualized sustainable dietary pattern (Phase 2: Weeks 13-20), and weight loss/remission maintenance (Phase 3: Weeks 21-52). We will determine if there is a preference for one diet over the other, measure satisfaction with each approach, and determine clinical outcomes (T2D remission, medication use, blood biomarkers) at one year. Qualitative interviews and feedback surveys with the participants, pharmacists, and RD will provide information on barriers and facilitators to each T2D remission strategy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-80 years old
* Diagnosed with T2D by a physician,
* HbA1c ≥ 6.0%,
* Body Mass Index ≥27 kg/m2 and
* No contraindications or dietary restrictions to following a low-carbohydrate/low-calorie diet.

Exclusion Criteria:

* History of heart disease, heart attack, heart failure, stroke or coronary artery disease within the previous 2 years,
* any current unstable cardiovascular disorder,
* history of liver disease,
* history of kidney disease with eGFR <30 mls/min/1.73 m2,
* history of neurological disease,
* previous bariatric surgery,
* weight loss (≥5%) within the last six months
* currently pregnant or lactating, or planning on becoming pregnant within the next 12 months,
* history of cancer within the previous 5 years,
* dietary restrictions or allergies that would inhibit adherence to the intervention diet,
* history of eating disorders,
* moderate or severe depression, anxiety or mental health condition that impacts daily life,
* currently following a low-carbohydrate or low-calorie diet, and
* unable to access the Internet (for communication with research team and RD).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Dual criteria for adherence to dietary interventions | 52 weeks
  defined as the proportion of participants attending ≥75% of visits with the pharmacist and/or registered dietitian (RD) and achieving at least 5% weight loss.
Intervention preference | 52 weeks
  the proportion of participants choosing each intervention
Type 2 diabetes remission | 52 weeks
  the proportion of participants achieving diabetes remission defined as Hemoglobin A1c (HbA1c) <6.5% and no glucose-lowering medications for at least 3 months, per international and new Canadian Clinical Practice Guidelines

SECONDARY OUTCOMES:
Body mass | weeks 0,12 ,20, 39, 52
  weight (kg) measured in-person for the LCal group and virtually for the LCarb group
Body mass index | weeks 0,12 ,20, 39, 52
  Calculated as kg/m2.
Waist circumference | weeks 0,12 ,20, 39, 52
  waist circumference (cm or in) measured in-person for the LCal group and virtually for the LCarb group
Blood pressure | weeks 0,12 ,20, 39, 52
  Average of two blood pressure measurements in-person for the LCal group and virtually for the LCarb group
Hemoglobin A1c | weeks 0,12 ,20, 39, 52
  Venous HbA1c (%) assessed in a clinical laboratory.
Fasting plasma glucose | weeks 0,12 ,20, 39, 52
  Fasting plasma glucose (mmol/L) assessed in a clinical laboratory.
Blood lipids | weeks 0,12 ,20, 39, 52
  Blood lipids (total cholesterol, high-density cholesterol, low-density cholesterol, triglycerides, non-HDL cholesterol, cholesterol/HDL ratio) assessed in a clinical laboratory.
Liver enzymes | weeks 0,12 ,20, 39, 52
  Liver enzymes (ALT, AST, GGT) assessed in a clinical laboratory.
C-reactive protein | weeks 0,12 ,20, 39, 52
  CRP (mg/L) assessed in a clinical laboratory.
Creatinine | weeks 0,12 ,20, 39, 52
  Creatinine (mg/dL) assessed in a clinical laboratory to infer glomerular filtration rate (GFR - mL/min).
Hematology panel (White blood cell count (WBC), Red blood cell count (RBC), Platelet count, Hematocrit red blood cell volume (HCT), Hemoglobin concentration (HB), Differential white blood count, Red blood cell indices. | weeks 0,12 ,20, 39, 52
  Hematology panel assessed in a clinical laboratory.
Hemoglobin A1c by finger pricks - only LCal group | weeks 0,12 ,20, 39, 52
  Capillary HbA1c (%) assessed in pharmacies by point-of-care equipment.
Diabetes medication | weeks 0,12 ,20, 39, 52
  Type and dosage of medication.
Anti-hypertensive medication | weeks 0,12 ,20, 39, 52
  Type and dosage of medication.
Physical activity questionnaire | weeks 0,12 ,20, 39, 52
  Physical activity will be assessed by the GODIN Questionnaire.
Sleep quality questionnaire | weeks 0,12 ,20, 39, 52
  Sleep will be assessed by the Pittsburg Sleep Quality Index (PSQI) questionnaire.
Hunger and satiety | weeks 0,12 ,20, 39, 52
  Hunger and satiety assessed by a hunger/fullness Visual Analogue Scale (VAS) questionnaire.
Quality of life | weeks 0,12 ,20, 39, 52
  Quality of life assessed by a self-rated health questionnaire (EQ-5D-5L).
2-hour postprandial hyperglycemia | weeks 0,12 ,20, 39, 52
  2-hour postprandial hyperglycemia measured by flash or continuous glucose monitoring for 14 days at each timepoint.
24hr average glucose area under the curve (AUC) | weeks 0,12 ,20, 39, 52
  24hr average glucose area under the curve (AUC) measured by flash or continuous glucose monitoring for 14 days at each timepoint.
Fasting glucose | weeks 0,12 ,20, 39, 52
  Fasting glucose measured by flash or continuous glucose monitoring for 14 days at each timepoint.
Glycemic variability | weeks 0,12 ,20, 39, 52
  Glycemic variability measured by flash or continuous glucose monitoring for 14 days at each timepoint.
Time in target range | weeks 0,12 ,20, 39, 52
  Time in target range measured by flash or continuous glucose monitoring for 14 days at each timepoint.
Glucose management indicator (GMI) | weeks 0,12 ,20, 39, 52
  Glucose management indicator (GMI) measured and calculated by flash or continuous glucose monitoring for 14 days at each timepoint.
Self-reported energy consumption | weeks 1,12 ,20, 39, 52
  Self-reported energy consumption will be assessed by 3-day food records at each timepoint.
Theory of planned behavior | weeks 0 and 52
  Theory of planned behavior assessed by • Theory of planned behavior (TPB) questionnaire.
Binge eating scale | weeks 0 and 52
  Binge eating scale assessed by a 16-item self-report questionnaire.
Self-esteem scale | weeks 0 and 52
  Self-esteem scale assessed by a 10-item scale questionnaire.
Diet Habit | weeks 0 and 52
  Diet habit assessed by a diet habit questionnaire.
Diet and food satisfaction | weeks 12 and 52
  Diet and food satisfaction assessed by a survey.
Preliminary economic analysis | week 52
  Assessed by costs of intervention against anticipated cost reductions based on medication use and health improvements (i.e. EQ-5D-5L);
Satisfaction, adherence and efficacy | week 52
  Satisfaction, adherence and efficacy will be assessed by a compilation of information: questionnaires, diet records, attendance to visits, weight loss, achievement of diabetes remission.
Feedback of the intervention with participants, RDs and pharmacists | week 52
  Feedback of the intervention through interviews/surveys with participants, RDs and pharmacists

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No